CLINICAL TRIAL: NCT00235820
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled Study Comparing the Safety and Efficacy of Adalimumab to Methotrexate in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Safety and Efficacy of Adalimumab to Methotrexate and Placebo in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: CHAMPION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Papierello/Director, Clinical Program Management, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M04-716
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; adalimumab
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: adalimumab
- B (Active Comparator)
  Interventions: Drug: MTX
- C (Placebo Comparator)
  Interventions: Drug: placebo adalimumab, placebo MTX

INTERVENTIONS:
Drug: adalimumab — 40 mg every other week following an 80 mg dose
  Other Names: ABT-D2E7; Humira
  Arms: A
Drug: MTX — MTX 7.5 to 25 mg once weekly
  Arms: B
Drug: placebo adalimumab, placebo MTX — placebo injections once every other week after 2 injections at Baseline (adalimumab) placebo capsules once weekly (MTX)
  Other Names: placebo
  Arms: C

SUMMARY:
Placebo-Controlled Study Comparing the Safety and Efficacy of Adalimumab to Methotrexate and Placebo in Subjects with Moderate to Severe Chronic Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in good health (Investigator discretion) with a recent stable medical history who has had a diagnosis of psoriasis for at least 12 months and stable moderate to severe chronic plaque psoriasis
* Subject is a candidate for systemic therapy or phototherapy and has active psoriasis despite treatment with topical agents.
* Subject was able and willing to self-administer sc injections or had available qualified person(s) to administer sc injections.
* Male subjects must hve been vasectomized or practicing birth control.

Exclusion Criteria:

* Previous systemic anti-TNF therapy.
* Prior use of MTX.
* Known hypersensitivity to the constituents of adalimumab.
* Systemic therapy for psoriasis for at least 4 weeks prior to Baseline; except for biologic therapies, which must be discontinued at least 12 weeks prior to enrollment.
* Topical psoriasis therapy for at least 2 weeks prior to Baseline, except for non-corticosteroid shampoos, bland (no alpha or beta hydroxy) emollients and low potency topical corticosteroids on the palms, soles, face, inframammary area, and groin only.
* Use of tanning beds, excessive sun exposure, or phototherapy (UVB, UVA), for at least 2 weeks prior to Baseline.
* Use of PUVA for at least 4 weeks prior to Baseline.
* Use of oral or injectable corticosteroids during the study.
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Female subject who is pregnant or breast feeding or considering becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2005-07; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving clinical response at Week 16 relative to the Baseline (Week 0) PASI score. | Week 16
Safety parameters | Every Study Visit

SECONDARY OUTCOMES:
Physician Global Assessment | Baseline - Week 16
PASI 50/90/100 | Baseline - Week 16
DLQI | Baseline - Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott
Locations (1):
- Global Medical Information-Abbott, Abbott Park, Illinois, United States

REFERENCES:
- [Derived] Papp KA, Armstrong AW, Reich K, Karunaratne M, Valdecantos W. Adalimumab Efficacy in Patients with Psoriasis Who Received or Did Not Respond to Prior Systemic Therapy: A Pooled Post Hoc Analysis of Results from Three Double-Blind, Placebo-Controlled Clinical Trials. Am J Clin Dermatol. 2016 Feb;17(1):79-86. doi: 10.1007/s40257-015-0161-5. PMID 26547918